CLINICAL TRIAL: NCT06243224
Title: The Effect Of High Intensity Interval Training And Moderate Intensity Continuous Training On Cardiopulmonary Parameters And Clinical Findings In Patients With Hypertension:A Randomized Comparative Study
Brief Title: The Effect Of High Intensity Interval Training And Moderate Intensity Continuous Training In Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nurdan Metin, Medical Doctor (Physical Medicine and Rehabilitation Resident Doctor), Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nurdan.mtn
Record Dates: First submitted 2024-01-13; First posted 2024-02-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Life Style
Keywords: Aerobic training; Hypertension; Aerobic capasity
MeSH Terms: conditions — Hypertension | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (HIIT) (Active Comparator): Patients will receive high intensity interval training (HIIT).
  Interventions: Other: High intensity interval training
- Moderate intensity (MICT) (Active Comparator): Patients will receive moderate intensity continuous training (MICT).
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: High intensity interval training — High intensity will be calculated based on load (watt) at % 75-85 of VO2 max analyzed during the CPET in HIIT group.Patients will perform 4 minutes of active high-intensity training with this load. Patients will perform for 1 minute each with a load (watt) of 50-60% of VO2 max in the interval phase.HIIT program will be performed with a horizontal ergometric bicycle (Ergoline GmbH ergoselect5, Serial no:2020010104, Germany ) for 3 sessions per week, each session being 30 minutes, for a total of 12 sessions for 4 weeks in the cardiopulmonary rehabilitation laboratory.
  Arms: High intensity interval training (HIIT)
Other: Moderate intensity continuous training — Moderate intensity will be calculated based on load (watt) at % 50-60 of VO2 max analyzed during the CPET in MICT group. Patients will complete their training sessions without changing this load determined during the treatment process.MICT program will be performed with a horizontal ergometric bicycle (Ergoline GmbH ergoselect5, Serial no:2020010104, Germany ) for 3 sessions per week, each session being 30 minutes, for a total of 12 sessions for 4 weeks in the cardiopulmonary rehabilitation laboratory.
  Arms: Moderate intensity (MICT)

SUMMARY:
Comparison of high intensity interval training (HIIT) and moderate intensity continuous training (MICT) in patients with hypertension patient in terms of aerobic capacity, blood pressure level, anxiety and depression scores, quality of life, kinesiophobia levels and sleep quality measurement.

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patients giving written informed consent will undergo screening period determine eligibility for study entry. The patients who met the eligibility recruitments will get into the assessment. The study will include 38 participants (19 HIIT and 19 MICT). Stratified randomization method will be preferred in this study.A total of 38 patients with primary hypertension will be included in the study to evaluate the effect of different intensities of aerobic exercise on cardiopulmonary parameters, aerobic capacity, blood pressure level, anxiety and depression scores, quality of life, kinesiophobia levels and sleep quality.The researcher will record demographic and clinical data of the patients.All patients will be randomly divided into two groups as MICT (n=19) and HIIT (n=19) group. All patients will be evaluated with BDI (Beck Depression Inventory), BAI (Beck Anxiety Inventory), SF-36 (Short Form-36), KCS (Kinesiophobia Causes Scalae), PSQI (Pittsburgh Sleep Quality Index) before starting the rehabilitation program. Cardiopulmonary exercise test (CPET) will be performed to analyze the cardiopulmonary parameters and determine exercise capacity of the patients.The exercise prescription will be tailored in two different intensities according to the VO2 max (maximum oxygen uptake) values of the patients (HIIT and MICT).For determination of exercise intensity, KPET will be applied to all patients using the Sentry Suite Version 2.19 program with the device (CareFusion Type Master Screen PFT, Serial no: 672819, Germany) at Ankara Bilkent City Hospital. Moderate intensity will be calculated based on load (watt) at % 50-60 of VO2 max, high intensity will be calculated based on load (watt) at % 75-85 of VO2 max analyzed during the CPET. The aerobic exercise program will be performed with a horizontal ergometric bicycle for 3 sessions per week, each session being 30 minutes, for a total of 12 sessions for 4 weeks in the cardiopulmonary rehabilitation laboratory. At the end of the rehabilitation program, all these parameters will be re-evaluated and analyzed in the two groups and the two groups will be compared in terms of these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Isolated Hypertension
* Being cognitively competent
* Being between the ages of 35-55
* Having given informed consent to participate in the study.

Exclusion Criteria:

* Clinical heart failure
* Uncontrolled hypertension
* Secondary hypertension
* Moderate or severe pulmoner disease
* Symptomatic peripheral arterial disease
* Unstable arrhythmia
* Unstable or severe angina
* Moderate or severe valvular heart disease
* Cognitive limitation unable to understand the research protocol
* Pace maker presence
* Language problem
* Autonomic neuropathy
* Cardiomyopathy
* Congenital heart disease
* Recent history of stroke
* Diabetes mellitus
* Severe musculoskeletal disease causing exercise limitation
* Being unable to continue treatment (3 days a week for 4 weeks)

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Aerobic capasity | baseline and at 4rd weeks
  The aim of this study was to demonstrate the effects of aerobic exercise on aerobic capacity in patients with hypertension.The primary outcome is the change in maksimum oxygen consumption (VO2 max: mL.kg-1.min-1) between baseline and week 4 measured during CPET. Aerobic capacity is a measure of the functional capacity of the cardiorespiratory system and can be expressed as VO2 max (ml O2/kg/min). VO2 max is the amount of oxygen consumed in milliliters per kilogram per minute. The most accurate and reliable measure of aerobic capacity is the measurement of maximum oxygen consumption (VO2 max), which is the maximum volume of oxygen the body can take up and use during exercise. An increase in VO2 max is the most reliable method of demonstrating the effect of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Metin, M.D, Principal Investigator — Ankara City Hospital Bilkent; Nilüfer Kutay Ordu Gökkaya, M.D, Study Director — Health Sciences University, Ankara Bilkent City Hospital; Ebru Alemdaroğlu, M.D, Study Chair — Health Sciences University, Ankara Bilkent City Hospital; Emre Aruğaslan, M.D, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Gorostegi-Anduaga I, Corres P, MartinezAguirre-Betolaza A, Perez-Asenjo J, Aispuru GR, Fryer SM, Maldonado-Martin S. Effects of different aerobic exercise programmes with nutritional intervention in sedentary adults with overweight/obesity and hypertension: EXERDIET-HTA study. Eur J Prev Cardiol. 2018 Mar;25(4):343-353. doi: 10.1177/2047487317749956. Epub 2018 Jan 9. PMID 29313359
- [Result] Ciolac EG, Bocchi EA, Bortolotto LA, Carvalho VO, Greve JM, Guimaraes GV. Effects of high-intensity aerobic interval training vs. moderate exercise on hemodynamic, metabolic and neuro-humoral abnormalities of young normotensive women at high familial risk for hypertension. Hypertens Res. 2010 Aug;33(8):836-43. doi: 10.1038/hr.2010.72. Epub 2010 May 7. PMID 20448634
- [Result] Williams B, Mancia G, Spiering W, Rosei EA, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I. [2018 ESC/ESH Guidelines for the management of arterial hypertension]. Kardiol Pol. 2019;77(2):71-159. doi: 10.5603/KP.2019.0018. No abstract available. Polish. PMID 30816983